CLINICAL TRIAL: NCT04388800
Title: Development of an Online Cognitive Behavioral Intervention Program to Reduce Depressive Symptoms for Hong Kong People With Depression
Brief Title: Online Cognitive Behavioral Intervention Program for Hong Kong People With Depression
Acronym: CANDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Stockholm University (Other); Richmond Fellowship of Hong Kong (Unknown); Caritas Wellness Link - Tsuen Wan (Unknown); Dr. Chiu Siu Ning (Unknown); Innovation and Technology Fund for Better Living (Unknown)
Responsible Party: Principal Investigator, Jiayan Pan, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITB/FBL/5002/18/P
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Depression
Keywords: online cognitive behavioral intervention; Hong Kong Chinese; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- web-based cognitive behavioral intervention (Experimental): The web-based program is consisted of 8 online modules, forum, internal messaging, reminder, online assessment and online booking. Each online module contains mood check, animation briefing and debriefing, case demonstration videos, session review and exercise.
  Blended mode is adopted to deliver service, which includes the online program, two face-to-face session and 2 telephone follow-ups with a clinical psychologist.
  Interventions: Other: Confront and Navigate Depression Online (CANDO)
- app-based cognitive behavioral intervention (Experimental): App-based cognitive behavioral intervention program The App-based program is consisted of 8 online modules, forum, internal messaging, reminder, online assessment and online booking. Each online module contains mood check, animation briefing and debriefing, case demonstration videos, session review and exercise.
  Blended mode is adopted to deliver service, which includes the online program, two face-to-face session and 2 telephone follow-ups with a clinical psychologist
  Interventions: Other: Confront and Navigate Depression Online (CANDO)
- Wait-list control group (No Intervention): No intervention will be provided when the experimental group is receiving services, but the access to the app-based program will be delivered to the wait-list control group after the two experimental groups complete the service.

INTERVENTIONS:
Other: Confront and Navigate Depression Online (CANDO) — This study adopts a blended mode of service delivery, which included both online and offline intervention. The online intervention includes 8 weekly online model, animation briefing and debriefing, case demonstration video, exercise, forum, internal messaging, reminder, online assessment, session review and online booking system. The offline intervention includes two face-to-face sessions and two telephone follow-ups.
  Arms: app-based cognitive behavioral intervention; web-based cognitive behavioral intervention

SUMMARY:
The purpose of this study is to develop a culturally and linguistically appropriate online cognitive behavioral intervention program-- with therapist guidance -- for Hong Kong Chinese adults suffering from major depressive disorder with mild to moderate depressive symptoms, and examine the effectiveness of this program in reducing their depressive symptoms and improving their mental health. The 3- and 6-month maintenance effect after 3 months and 6 months will also be tested.

DETAILED DESCRIPTION:
Previous studies have demonstrated that online cognitive behavioral therapy can significantly reduce depressive symptoms and improve mental health for people with depression. This project will develop an online cognitive behavioral intervention program (including both an online platform and a smartphone application) for Hong Kong people with depression. Blended mode will be delivered service, which include 8-week online program, 2 face-to-face sessions and 2 telephone follow-ups by a clinical psychologist. The program will be evaluated in its effectiveness in reducing depressive and anxiety symptoms, psychological distress, negative thoughts and negative emotions and increasing positive thoughts and positive emotions.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong resident
* Has mild to moderate depressive symptoms
* No suicidal risk in the past 3 months
* Receive no face-to-face counselling since program commencement
* Has access to a computer/smartphone with internet access
* Has a valid email address

Exclusion criteria:

* Has severe or no depressive symptoms
* Has suicidal risk in the past 3 months
* Currently receiving other psychological treatment
* Suffer from severe psychiatric conditions, such as bipolar disorder or schizophrenia
* Has no computer or smartphone with internet access
* Has no valid email address

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | 6 months
  21-item rating scale for depressive symptoms
Patient Health Questionnaire-9 (PHQ-9) | 6 months
  9-item rating scale for depressive symptoms.

SECONDARY OUTCOMES:
General Health Questionnaire-12 (GHQ-12) | 6 months
  12 item rating scale for psychological distress.
Beck Anxiety Inventory (BAI) | 6 months
  21-item rating scale for symptoms of anxiety.
Chinese Automatic Thoughts Questionnaire (CATQ) | 6 months
  20-item rating scale for automatic thoughts.
Chinese Affect Scale (CAS) | 6 months
  20-item rating scale for positive and negative emotions of Chinese-speaking people.
Negative effects Questionnaire (NEQ) (administered at post-test only) | 6 months
  20-item rating scale for negative effects caused by psychological treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Jiayan Pan, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pan JY, Rafi J. Culturally Adapted Guided Internet-Based Cognitive Behavioral Therapy for Hong Kong People With Depressive Symptoms: Randomized Controlled Trial. J Med Internet Res. 2025 Feb 25;27:e64303. doi: 10.2196/64303. PMID 39998865